CLINICAL TRIAL: NCT06854627
Title: Effect of Continuous Prolonged Prone Position Versus Intermittent Daily Prone Position on Mortality in ARDS Patients: A Multicenter Randomized Controlled Trial
Brief Title: Effect of Continuous Prolonged Prone Position Versus Intermittent Daily Prone Position in ARDS
Acronym: ePRONE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Collaborators: Hospital do Coracao (Other); Fundacion Clinica Valle del Lili (Other); Fondo Nacional de Desarrollo Científico y Tecnológico, Chile (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 230606007
Record Dates: First submitted 2025-01-21; First posted 2025-03-03 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-04

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: ACUTE RESPIRATORY DISTRESS SYNDROME; RESPIRATORY FAILURE; PRONE POSITION; MECHANICAL VENTILATION
MeSH Terms: conditions — Respiratory Distress Syndrome; Respiratory Insufficiency

STUDY DESIGN:
Intervention Model Description: Study do not use Drug, Biological/Vaccine, or Combination Product.
Who Masked: Outcomes Assessor
Masking Description: groups will be coded for the assessment of the outcomes
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intermittent Prone Position (Active Comparator): This arm will receive prone position sessions as applied in the PROSEVA trial (Guerin 2013)
  Interventions: Procedure: Daily prone position sessions
- Prolonged Prone Position (Experimental): This arm will receive prone position sessions as applied in a previous multicenter study during the COVID-19 pandemics (Cornejo 2022)
  Interventions: Procedure: Prolonged prone position sessions

INTERVENTIONS:
Procedure: Daily prone position sessions — Prone position sessions will be extended at least 16 hours, but no longer than 24 hours. Prone sessions will be repeated if PaO2/FiO2 ratio decreases to < 150 after returning to supine position within the first 7 days after randomization. The extension of repeated prone sessions will follow the same criteria.
  Arms: Intermittent Prone Position
Procedure: Prolonged prone position sessions — Prone position sessions will be extended at least 48 hours AND until PaO2/FiO2 ratio is ≥ 200, but no longer than 120 hours. Prone sessions will be repeated if PaO2/FiO2 ratio decreases to < 150 after returning to supine position within the first 7 days after randomization. The extension of repeated prone sessions will follow the same criteria.
  Arms: Prolonged Prone Position

SUMMARY:
Prone position (placing the patient on his abdomen) has been shown to be an effective intervention to decrease mortality in adults connected to mechanical ventilation for moderate to severe Acute Respiratory Distress Syndrome (ARDS). Patients may require one or more sessions of prone position. However, the optimal duration of prone sessions is unknown. The goal of this clinical trial is to learn if applying prone position in prolonged sessions (> 48 hours - prolonged prone position) is more effective than applying it in daily sessions (16 to 24 hours - intermittent prone position). The trial will also learn about the safety of prolonged prone position compared to intermittent prone position. The main questions it aims to answer are:

* Does prolonged prone position increase survival compared to intermittent prone position in participants with moderate to severe ARDS ?
* How does prolonged prone position compare to intermittent prone position in terms of medical problems associated to prone position ?

Researchers will compare prolonged versus intermittent prone position to see which approach is better to treat moderate to severe ARDS.

Participants will:

* Receive prone position either in prolonged (> 48 hours) or daily (16 to 24 hours) sessions during the first 7 days
* Be followed for up to 90 days to assess their clinical evolution

DETAILED DESCRIPTION:
Acute Respiratory Distress Syndrome (ARDS) is a severe condition with a 40% mortality rate. The management of ARDS still relies largely on supportive therapy. The cornerstone of this support is protective mechanical ventilation to prevent ventilator-induced lung injury (VILI). For patients with moderate-to- severe forms of ARDS, specifically mechanically ventilated patients with PaO2/FiO2 ratios below 150, the use of prone position has shown to be a fundamental intervention which became one of the most relevant pillars of the ICU management during the Covid-19 pandemics. Several studies have shown that prone position not only improves oxygenation, but can attenuate the mechanisms of VILI, which would explain its benefit in terms of mortality. The physiologic benefits of prone position are progressive along time, but they can be lost rapidly after returning to supìne position.

Since the publication of the landmark PROSEVA study (Guerin 2013), which showed that ventilating patients in prone position decreased mortality, the standard approach to prone position has been the use of daily sessions of 16 to 20 hours. With this approach most patients usually require 3 to 4 prone sessions (intermittent daily prone position). However, due to the excessive workload of ICU staff during the Covid-19 pandemics, several centers decided to extend the sessions beyond 24 hours to decrease the frequency of position changes in patients with Covid-19 associated ARDS. Several centers reported their experience with prolonged sessions showing that it was feasible and that the rate of adverse events appeared to be similar to those previously reported with the standard daily sessions. The largest experience reported up to now was a retrospective study which included 417 patients from 15 centers in Chile, where a continuous prolonged prone position was applied as a nationwide strategy (Cornejo 2022). Most patients required a single prone session of 4 (3-5) days. Although the study lacked a control group, the mortality and rate of adverse events was rather low compared to other series of patients with similar characteristics. A non-randomized controlled study from 3 hospital in US even showed that compared to patients treated with standard prone sessions (< 24 hours), patients treated with prolonged sessions had a lower risk of mortality (Okin 2023). However, other reports have shown conflicting results regarding the potential benefit associated to prolonging prone position sessions beyond 24 hours. Recent guidelines have acknowledged that the optimal duration of prone position sessions is unknown and must be further investigated (Grasselli 2023). Prolonging prone position sessions may ensure that this lung protective intervention is maintained throughout the acute phase of ARDS.

The goal of the present study is to compare the effects of a continuous prolonged prone position versus an intermittent daily prone position on mortality and other relevant outcomes, as well as on the incidence of adverse events potentially related to prone position, in mechanically ventilated patients with moderate-to-severe ARDS.

The study will be a randomized, multicenter, two-arm parallel-group, investigator-led clinical trial with allocation concealment and intention-to-treat analysis. Patients allocated to the experimental arm (prolonged prone position) will receive prone position sessions for a minimum of 48 hours, which will be further extended until PaO2/FiO2 is ≥ 200, or until reaching the maximum of 120 hours. Patients allocated to the control arm (intermittent prone position) will receive prone position sessions for a minimum of 16 hours and a maximum of 24 hours. In both groups prone sessions may be repeated if PaO2/FiO2 ratio falls below 150 after being returned to supine position during the first 7 days (intervention period).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Endotracheal intubation and mechanical ventilation for less than 72 hours
* Moderate-severe ARDS defined as:

  1. Within 1 week of a known clinical insult or new or worsening respiratory symptoms
  2. Bilateral infiltrates not fully explained by effusions, lobar/lung collapse, or nodules
  3. Respiratory failure not fully explained by cardiac failure or fluid overload
  4. PaO2/FiO2 < 150 mmHg in supine position
* Prone positioning has been indicated by the attending physician, OR has already been initiated within the last 16 hours

Exclusion Criteria:

* Contraindications for prone positioning such as intracranial pressure > 20 mmHg, massive hemoptysis, recent tracheal surgery or sternotomy or abdominal surgery with an open wound, recent facial trauma or facial surgery, unstable spine, femur, or pelvic fractures, or a single anterior chest tube with air leaks
* Patient on extracorporeal membrane oxygenation (ECMO) before randomization
* Chronic respiratory failure requiring oxygen therapy or non-invasive ventilation (NIV)
* Known pregnancy
* Anticipating withdrawal of life support or shift to palliative care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 780 (Estimated)
Dates: Start 2025-04-07 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
28-day mortality | 28 days
  All-cause mortality

SECONDARY OUTCOMES:
90-day mortality | 90 days
  All-cause mortality
Ventilator-free days | 28 days
  Days-free from mechanical ventilation and alive up to day 28
Hospital-free days at day 28 | 28 days
  Days-free from Hospital and alive up to day 28

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro Bruhn, MD, PhD, Principal Investigator — Pontifiia Universidad Catolica de Chile; Rodrigo Cornejo, MD, MBA, Study Director — University of Chile
Locations (6):
- Chile (6):
  - Hospital Guillermo Grant Benavente, Concepción
  - Complejo Asistencial Dr. Victor Ríos Ruiz, Los Ángeles
  - Hospital de Quilpué, Quilpué
  - Clínica Las Condes, Santiago
  - Hospital Clínico UC Christus, Santiago
  - Hospital Clínico Universidad de Chile, Santiago

IPD SHARING:
Plan to Share IPD: Yes
anonymized data will be shared among reasonable request to the corresponding author.
Supporting Information: Study Protocol, SAP
Time Frame: will become available after the main paper is published, for 10 years.
Access Criteria: among reasonable request to the principal investigator

REFERENCES:
- [Background] Cornejo RA, Montoya J, Gajardo AIJ, Graf J, Alegria L, Baghetti R, Irarrazaval A, Santis C, Pavez N, Leighton S, Tomicic V, Morales D, Ruiz C, Navarrete P, Vargas P, Galvez R, Espinosa V, Lazo M, Perez-Araos RA, Garay O, Sepulveda P, Martinez E, Bruhn A; SOCHIMI Prone-COVID-19 Group. Continuous prolonged prone positioning in COVID-19-related ARDS: a multicenter cohort study from Chile. Ann Intensive Care. 2022 Nov 28;12(1):109. doi: 10.1186/s13613-022-01082-w. PMID 36441352
- [Background] Guerin C, Reignier J, Richard JC, Beuret P, Gacouin A, Boulain T, Mercier E, Badet M, Mercat A, Baudin O, Clavel M, Chatellier D, Jaber S, Rosselli S, Mancebo J, Sirodot M, Hilbert G, Bengler C, Richecoeur J, Gainnier M, Bayle F, Bourdin G, Leray V, Girard R, Baboi L, Ayzac L; PROSEVA Study Group. Prone positioning in severe acute respiratory distress syndrome. N Engl J Med. 2013 Jun 6;368(23):2159-68. doi: 10.1056/NEJMoa1214103. Epub 2013 May 20. PMID 23688302
- [Background] Grasselli G, Calfee CS, Camporota L, Poole D, Amato MBP, Antonelli M, Arabi YM, Baroncelli F, Beitler JR, Bellani G, Bellingan G, Blackwood B, Bos LDJ, Brochard L, Brodie D, Burns KEA, Combes A, D'Arrigo S, De Backer D, Demoule A, Einav S, Fan E, Ferguson ND, Frat JP, Gattinoni L, Guerin C, Herridge MS, Hodgson C, Hough CL, Jaber S, Juffermans NP, Karagiannidis C, Kesecioglu J, Kwizera A, Laffey JG, Mancebo J, Matthay MA, McAuley DF, Mercat A, Meyer NJ, Moss M, Munshi L, Myatra SN, Ng Gong M, Papazian L, Patel BK, Pellegrini M, Perner A, Pesenti A, Piquilloud L, Qiu H, Ranieri MV, Riviello E, Slutsky AS, Stapleton RD, Summers C, Thompson TB, Valente Barbas CS, Villar J, Ware LB, Weiss B, Zampieri FG, Azoulay E, Cecconi M; European Society of Intensive Care Medicine Taskforce on ARDS. ESICM guidelines on acute respiratory distress syndrome: definition, phenotyping and respiratory support strategies. Intensive Care Med. 2023 Jul;49(7):727-759. doi: 10.1007/s00134-023-07050-7. Epub 2023 Jun 16. PMID 37326646
- [Background] Okin D, Huang CY, Alba GA, Jesudasen SJ, Dandawate NA, Gavralidis A, Chang LL, Moin EE, Ahmad I, Witkin AS, Hardin CC, Hibbert KA, Kadar A, Gordan PL, Lee H, Thompson BT, Bebell LM, Lai PS. Prolonged Prone Position Ventilation Is Associated With Reduced Mortality in Intubated COVID-19 Patients. Chest. 2023 Mar;163(3):533-542. doi: 10.1016/j.chest.2022.10.034. Epub 2022 Nov 4. PMID 36343687